CLINICAL TRIAL: NCT06666686
Title: The Effect of Noise Control During Anesthesia Induction in Laparoscopic Cholecystectomy Surgery on Postoperative Hemodynamic Parameters, Pain, Nausea and Vomiting, and Recovery Time From Anesthesia
Brief Title: The Effect of Noise Control During Anesthesia Induction in Laparoscopic Cholecystectomy Surgery
Acronym: Anesth-noise
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Cagla AVCU, Research Assistant, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Anesthesia noise
Record Dates: First submitted 2024-10-19; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cholecystectomy, Laparoscopic; Noise; Anesthesia Induction
Keywords: Anesthesia induction; Noise control; Laparoscopic cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Control group
- Active noise control (Experimental): This is the group where active noise control headphones are applied. Headphones will be applied to patients from the beginning to the end of anesthesia induction.
  Interventions: Device: Active noise control headphone
- Passive noise control (Experimental): This is the group where passive noise control headphones are applied. Headphones will be applied to patients from the beginning to the end of anesthesia induction.
  Interventions: Device: Passive noise control headphone

INTERVENTIONS:
Device: Active noise control headphone — This is the group where active noise control headphones are applied. Headphones will be applied to patients from the beginning to the end of anesthesia induction.
  Arms: Active noise control
Device: Passive noise control headphone — This is the group where passive noise control headphones are applied. Headphones will be applied to patients from the beginning to the end of anesthesia induction.
  Arms: Passive noise control

SUMMARY:
This study aims to determine the effects of active and passive noise control method and headphone usage and noise level during anesthesia induction in laparoscopic cholecystectomy surgery on hemodynamic parameters, pain, nausea and vomiting, and recovery time from anesthesia in patients after surgery.

DETAILED DESCRIPTION:
When the studies in the literature are examined, there is no study evaluating the effects of noise level and active and passive noise control method and headphone usage during anesthesia induction on patients undergoing laparoscopic cholecystectomy surgery, which is the most frequently applied among laparoscopic surgeries.

This study aims to eliminate these deficiencies in the literature, to reveal the benefits of active and passive noise control headphone usage for noise control as it is an easy and cheap method and has no side effects, and to popularize this application.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-65,
* Diagnosed with cholecystitis or cholelithiasis,
* Planned for elective laparoscopic cholecystectomy,
* Have an ASA I or ASA II anesthesia classification,
* Oriented to person, place and time,
* Undergoing general anesthesia,
* Not having a psychiatric or cognitive/mental disease (dementia etc.),
* Not having vision, hearing and communication problems,
* Speaking, reading and writing Turkish,
* Patients who agree to participate in the study verbally and in writing will be included.

Exclusion Criteria:

* Patients who underwent spinal anesthesia,
* Transferred to units such as intensive care after surgery,
* Underwent emergency laparoscopic cholecystectomy,
* Patients who were planned for elective open cholecystectomy will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Identification Form | Pre-intervention
  This form, prepared by researchers in line with the literature, consists of questions about the individual and surgical characteristics of the patients.
Patient Follow-up Form-Part 1 | perioperative
  This part includes the evaluation and recording of the patients' hemodynamic parameters (temperature (°C), pulse rate(dk), respiratory rate (dk), oxygen saturation (%) and blood pressure (mmHg)) after admission to the operating room, during the anesthesia induction phase, during the surgical process from the end of anesthesia induction to the termination of anesthesia and every 15 minutes in the post-anesthesia care unit.
Patient Follow-up Form-Part-2 | before surgery (anesthesia induction phase)
  In this part, the noise level measurement during the anesthesia induction phase will be recorded.
Patient Follow-up Form-Part-3 (Numerical Analog Scale) | in the post-anesthesia care unit (up to 2 hours post surgery)
  This part is used to measure the pain intensity of patients in the post-anesthesia care unit. The form consists of a 10 cm long ruler with pain intensity scores ranging from 0 to 10, with "0 = No Pain" and "10 = Most Severe Pain".
Patient Follow-up Form-Part-4 (Visual Analog Scale for Assessment of Nausea) | in the post-anesthesia care unit (up to 2 hours post surgery)
  This scale is used to measure the severity of nausea in patients in the post-anesthesia care unit. The severity of nausea is scored by the patient between 0 and 10 using a 100 mm long ruler, with "0 = No Nausea at All" and "100 = Most Severe Nausea Possible".
Patient Follow-up Form-Part-5 (Modified Aldrete Score) | in the post-anesthesia care unit (up to 2 hours post surgery)
  It is a scoring system used to assess whether patients are ready to be transferred from the post-anesthesia care unit to the clinic. It consists of 5 parameters: "Activity", "Respiration", "Circulation", "Consciousness" and "Oxygen Saturation" and each parameter is scored as "0", "1" and "2". A total score of 9 and above indicates that transfer to the clinic is appropriate.
Patient Follow-up Form-Part-6 | in the post-anesthesia care unit (up to 2 hours post surgery)
  The part includes the vomiting (if any, how many times), status of premedication, anesthetic drugs, anesthesia induction duration, the duration between anesthesia induction and the termination of anesthesia, and the duration of stay in the post-anesthesia care unit.
Noise Meter | before surgery (anesthesia induction phase)
  During the anesthesia induction phase, the noise level of the operating room will be measured with a handheld noise measuring device. The device will be placed approximately 120 cm away from the patient's head. The noise level will be measured and recorded from the beginning of anesthesia induction to termination.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Namık Kemal University, Tekirdağ, Suleymanpasa
  - Namık Kemal University, Tekirdağ, Süleymanpaşa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] You S, Xu F, Zhu X, Qin S, Zheng X, Tao C, Wu Y, Chen Y, Shu B, Huang H, Duan G. Effect of intraoperative noise on postoperative pain in surgery patients under general anesthesia: evidence from a prospective study and mouse model. Int J Surg. 2023 Dec 1;109(12):3872-3882. doi: 10.1097/JS9.0000000000000672. PMID 37598384
- [Background] You S, Xu F, Wu Y, Qin S, Shu B, Chen Y, Chen Y, Huang H, Duan G. Effect of noise isolation using noise-cancelling headphones during laparoscopic surgery for postoperative pain reduction: A randomized clinical trial. J Clin Anesth. 2024 Feb;92:111286. doi: 10.1016/j.jclinane.2023.111286. Epub 2023 Oct 12. PMID 37837796
- [Background] Belyad S, Talakoub R, Aarabi A. The Effect of Soundproof Headphones During Orthopedic Surgery Under Spinal Anesthesia on Patients' Physiological Indices and Duration of Recovery: A Randomized, Controlled, Clinical Trial. J Perianesth Nurs. 2024 Jun;39(3):379-385. doi: 10.1016/j.jopan.2023.08.016. Epub 2024 Jan 4. PMID 38180393